CLINICAL TRIAL: NCT00800748
Title: An Open, Phase IV, Multicentric Study, Evaluating Safety and Efficacy of Ribavirin (Copegus®) and Peginterferon Alfa-2a (Pegasys®) Combination in Specific Groups
Brief Title: A Study of Combination Treatment With Peginterferon Alfa-2a (Pegasys) Plus Ribavirin (Copegus) in Participants With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19387; 2005-003932-23 (EudraCT Number)
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Participants with genotype 1, 4, 5 or 6 received peginterferon alfa-2a 180 mcg SC qw + ribavirin 1000-1200 mg PO daily (dependent on body weight) for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Group B (Experimental): Participants with genotype 2 or 3 received peginterferon alfa-2a 180 mcg SC qw + ribavirin 800 mg PO daily for 24 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Group C (Experimental): Participants with HIV co-infection received peginterferon alfa-2a 180 mcg SC qw + ribavirin 800 mg PO daily for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a was administered at a dose of 180 mcg SC weekly for 48 weeks to participants with genotype 1, 4, 5, 6 and to participants with HIV co-infection, or for 24 weeks to participants with genotype 2 and 3.
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin was administered at a dose of 1000-1200 mg PO daily for 48 weeks to participants with genotype 1, 4, 5, 6 or 800 mg PO daily for 24 weeks to participants with genotype 2 and 3.
  Other Names: Copegus

SUMMARY:
This 3-arm study assessed the safety and efficacy of combination treatment with peginterferon alfa-2a + ribavirin in participants with chronic hepatitis C. Three groups of participants were studied; 1) those with elevated alanine transaminase (ALT) levels, 2) those with normal ALT levels, and 3) those with human immunodeficiency virus (HIV) co-infection. Participants with genotype 1, 4, 5 or 6 received peginterferon alfa-2a 180 micrograms (mcg) subcutaneous (SC) once weekly (qw) + ribavirin 1000-1200 milligrams (mg) orally (PO) daily (dependent on body weight) for 48 weeks. Those with genotype 2 or 3 received peginterferon alfa-2a 180 mcg SC qw + ribavirin 800 mg PO daily for 24 weeks, and all participants with HIV co-infection received peginterferon alfa-2a 180 mcg SC qw + ribavirin 800 mg PO daily for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants at least 18 years of age
* Chronic hepatitis C, with detectable serum hepatitis C virus (HCV) ribonucleic acid (RNA)
* Scheduled for treatment with peginterferon alfa-2a
* Compensated liver disease
* Women in fertile age must be informed about obligation of using adequate contraception during and 6 months post treatment with ribavirin (Copegus®)
* Men with a sexual partner in fertile age must be informed about obligatory contraception preventing pregnancy during the course of treatment with ribavirin (Copegus®) as well as 6 months after treatment cessation
* Female participants in the study must have a negative pregnancy test performed not sooner than within 2 weeks preceding the planned inclusion to the study
* Men with a sexual partner in fertile age must produce a negative result of the partner's pregnancy test performed not sooner than within 2 weeks preceding the planned partner's inclusion to the study

Exclusion Criteria:

* Chronic liver disease other than chronic hepatitis C
* Active hepatitis A virus or hepatitis B virus infection
* Therapy with any systemic antiviral, antineoplastic or immunomodulatory treatment less than or equal to (<=) 6 months prior to first dose of study drug
* Hemoglobin <120 grams per liter (g/L) in female participants or <130 g/L in male participants (the result must not be older than 2 weeks prior to inclusion to the study)
* Platelet count <90 x 10^9/liter (the result must not be older than 2 weeks prior to inclusion to the study
* Neutrofil count <1.5 x 10^9/liter (the result must not be older than 2 weeks prior to inclusion to the study)
* Participants with increased risk of anaemia, or participants at risk of serious health problems resulting from anaemia or decrease of hemoglobin (e.g., participants with serious cardiovascular or cerebrovascular disease)
* History or presence of a serious mental disease, especially depression, which, in the investigator's opinion, does not allow administration of peginterferon alfa-2a (Pegasys®)
* History or presence of a disease consequent to immunodeficiency (e.g., inflammatory diseases of intestine, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, rheumatoid arthritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2006-02-01 (Actual); Primary Completion 2009-01-09 (Actual); Study Completion 2009-01-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virological Response | Up to 72 weeks
  Sustained virological response is defined as having no hepatitis C (HCV) virus detectable in the blood 24 weeks after end of treatment.

SECONDARY OUTCOMES:
Percentage of Participants With End-of-Treatment Virological Response | Up to 48 weeks
  End-of-treatment virological response is defined as having no HCV virus detectable in the blood immediately after end of treatment.
Percentage of Participants With Early-Treatment Virological Response | Up to 12 weeks
  Early-treatment virological response is defined as having no HCV virus detectable in the blood or a 2-log (100-fold) decrease in HCV virus concentration in the blood after 12 weeks of study treatment.
Percentage of Participants With Adverse Events | Up to 72 weeks
  An adverse event is considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsen during the study are reported as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- Czechia (23):
  - Beroun
  - Brno
  - Chomutov
  - Česká Lípa
  - České Budějovice
  - Děčín
  - Havířov
  - Havlíčkův Brod
  - Hradec Králové
  - Jablonec/nisou
  - Jihlava
  - Karlovy Vary
  - Kolín
  - Liberec
  - Mělník
  - Most
  - Olomouc
  - Opava
  - Ostrava
  - Pardubice
  - Prague
  - Prostějov
  - Ústí nad Labem
- Slovakia (5):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Martin
  - Trenčín